CLINICAL TRIAL: NCT07178821
Title: Sling-Fiber Preservation POEM vs. Conventional POEM for Reducing Post-POEM GERD: A Randomized Control Trial
Brief Title: Sling-Fiber Preservation POEM vs. Conventional POEM for Reducing Post-POEM GERD
Acronym: SFP-POEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Hoag Memorial Hospital Presbyterian (Other); University of Ottawa (Other); Vancouver General Hospital (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Frances Dang, Assistant Clinical Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7028
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Achalasia, Esophageal; GERD (Gastroesophageal Reflux Disease)
Keywords: Achalasia; POEM; Peroral Endoscopic Myotomy; Sling Fiber Preservation; SFP-POEM; Gastroesophageal Reflux; GERD; Reflux Esophagitis; Randomized Controlled Trial
MeSH Terms: conditions — Esophageal Achalasia; Gastroesophageal Reflux; Esophagitis, Peptic

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1 ratio to receive either sling fiber-preservation POEM or conventional POEM. Each participant undergoes only one assigned intervention and is followed for 12 months.
Who Masked: Participant
Masking Description: Participants are blinded to the intervention group. Endoscopists performing the procedure cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional POEM (Active Comparator): Participants in this arm will undergo standard peroral endoscopic myotomy (POEM), including myotomy of circular and sling muscle fibers at the gastric side.
  Interventions: Procedure: Conventional POEM
- Sling Fiber-Preservation POEM (Experimental): Participants in this arm will undergo posterior POEM with selective preservation of the gastric sling fibers. Myotomy is performed to the right of the second penetrating vessel to spare the sling fibers. The double scope technique will be employed to confirm that the tunnel ends on the lesser curve, which confirms sparing of the sling fibers.
  Interventions: Procedure: Sling Fiber-Preserving POEM

INTERVENTIONS:
Procedure: Conventional POEM — Standard posterior POEM with full-thickness myotomy, including both circular and gastric sling muscle fibers.
  Arms: Conventional POEM
Procedure: Sling Fiber-Preserving POEM — Posterior POEM with selective preservation of gastric sling fibers by limiting myotomy to the right of the second penetrating vessel.
  Other Names: SFP-POEM
  Arms: Sling Fiber-Preservation POEM

SUMMARY:
Peroral endoscopic myotomy (POEM) is an effective, minimally invasive treatment for achalasia, offering excellent rates of symptom relief. However, a significant drawback is the high incidence of gastroesophageal reflux disease (GERD) following the procedure. One proposed technical modification, the selective preservation of the sling fibers during gastric myotomy (SFP-POEM), may reduce this risk without compromising efficacy as compared to a conventional POEM procedure, which includes myotomy of the sling fibers. In this study, adults with achalasia will be randomly assigned to receive one of the two POEM technical approaches. Researchers will monitor whether preserving sling fibers reduces the rates of reflux esophagitis (classified as Los Angeles Grade B or higher) on follow-up endoscopy. Participants will be followed for up to 1 year after the procedure.

DETAILED DESCRIPTION:
Achalasia is a rare esophageal motility disorder treated effectively with peroral endoscopic myotomy (POEM). However, post-procedure gastroesophageal reflux disease (GERD) is a common complication, reported in up to 65% of cases. One proposed technical modification - the selective preservation of gastric sling fibers - may help reduce reflux by maintaining part of the native anti-reflux mechanism.

This is a single-blinded, multicenter randomized controlled trial comparing sling fiber preservation (SFP) POEM versus conventional POEM in adult patients with achalasia. Patients are randomized 1:1 to either technique. The primary endpoint is the incidence of significant reflux esophagitis (LA esophagitis grade B or higher) at 3 months post-procedure endoscopy. Secondary outcomes include acid exposure time on pH impedence monitoring, symptomatic reflux (GerdQ), PPI usage, technical and clinical success, and adverse events. Follow-up continues for 12 months.

The study aims to determine whether the SFP-POEM technique reduces acid reflux without compromising treatment efficacy.

ELIGIBILITY:
Inclusion Criteria (Participants must meet all of the following):

* Age ≥ 18 years
* Diagnosis of achalasia (Type I-III) per Chicago Classification v3.0
* Deemed appropriate candidates for POEM
* Ability to provide informed consent

Exclusion Criteria (Participants will be excluded if any of the following apply):

* Spastic motility disorders other than achalasia type I-III (e.g. diffuse esophageal spasm, jackhammer esophagus, EGJ outflow obstruction)
* Sigmoid esophagus
* Prior surgical myotomy (e.g., Heller myotomy)
* Contraindications to endoscopy or general anesthesia
* Pregnancy or actively breastfeeding
* Significant cardiopulmonary comorbidities that preclude safe endoscopic intervention
* Coagulopathy or portal hypertension
* Unwillingness or inability to complete follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Significant Reflux Esophagitis (Los Angeles Grade B or Higher) | 3 months post-procedure
  Reflux esophagitis will be assessed by upper endoscopy (EGD) at 3 months post-POEM. Grading will be based on the Los Angeles (LA) Classification. Significant reflux is defined as LA Grade B or higher.

SECONDARY OUTCOMES:
Esophageal Acid Exposure | 3 months post-procedure
  Esophageal acid exposure will be measured by 24-hour Bravo pH monitoring performed off PPIs for at least 2 weeks. Reflux severity is quantified using acid exposure time (%) and the DeMeester composite score. The DeMeester score has no fixed maximum; higher values indicate greater esophageal acid exposure. Pathologic reflux is defined as acid exposure time >6% and/or a DeMeester score >14.72.
Symptomatic Gastroesophageal Reflux (GerdQ Score) | 3, 6, 12 months post-procedure
  Symptom-based GERD assessment will be measured using the Gastroesophageal Reflux Disease Questionnaire (GerdQ), which ranges from 0 to 18. Higher scores indicate more frequent or severe reflux symptoms, while lower scores indicate fewer or no symptoms. A score >7 is considered clinically significant.
Proton Pump Inhibitor (PPI) Use | 3, 6, 12 months post-procedure
  Assessment of ongoing PPI therapy and symptom-guided discontinuation based on reflux control.
Clinical Success (Eckardt Symptom Score ≤ 3) | 3, 6 and 12 months post-procedure
  Symptom improvement will be measured using the Eckardt Symptom Score, which ranges from 0 to 12. Higher scores indicate more severe symptoms (dysphagia, chest pain, regurgitation, and weight loss), while lower scores indicate symptom improvement. A score ≤ 3 is considered a successful clinical outcome.
Technical Success | During procedure
  Technical success defined as completion of full-length myotomy as planned.
Adverse Events | Within 1 month post-procedure
  Monitoring of intra- and post-procedural complications, including bleeding, perforation, capno-peritoneum, leak, infection, and other unexpected events.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Samarasena, MD, MBA, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine - UCI Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared outside the study team. The current protocol does not include provisions for public or external data sharing.

REFERENCES:
- [Background] Nabi Z, Chandran V, Basha J, Ramchandani M, Inavolu P, Kalpala R, Goud R, Jagtap N, Darisetty S, Gupta R, Tandan M, Lakhtakia S, Kotla R, Devarasetty R, Rao GV, Reddy DN. Conventional versus oblique fiber-sparing endoscopic myotomy for achalasia cardia: a randomized controlled trial (with videos). Gastrointest Endosc. 2024 Jan;99(1):1-9. doi: 10.1016/j.gie.2023.08.007. Epub 2023 Aug 19. PMID 37598863
- [Background] Fujiyoshi Y, Fujiyoshi MRA, Khalaf K, May GR, Teshima CW. Sling fiber preservation during POEM reduces incidence of postoperative reflux symptoms. Dis Esophagus. 2025 Jan 7;38(1):doae097. doi: 10.1093/dote/doae097. PMID 39586589
- [Background] Tanaka S, Toyonaga T, Kawara F, Watanabe D, Hoshi N, Abe H, Ariyoshi R, Ohara Y, Takao T, Morita Y, Umegaki E, Kodama Y. Novel per-oral endoscopic myotomy method preserving oblique muscle using two penetrating vessels as anatomic landmarks reduces postoperative gastroesophageal reflux. J Gastroenterol Hepatol. 2019 Dec;34(12):2158-2163. doi: 10.1111/jgh.14814. Epub 2019 Aug 23. PMID 31373050
- [Background] Shiwaku H, Inoue H, Shiwaku A, Okada H, Hasegawa S. Safety and effectiveness of sling fiber preservation POEM to reduce severe post-procedural erosive esophagitis. Surg Endosc. 2022 Jun;36(6):4255-4264. doi: 10.1007/s00464-021-08763-w. Epub 2021 Oct 29. PMID 34716481